CLINICAL TRIAL: NCT03024814
Title: Prophylactic Acetaminophen for Prevention Intraventricular Hemorrhage in Premature Infants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Mountasser Al-Mouqdad, NICU consultant, King Saud Medical City
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HRC-09-Nov15-02
Record Dates: First submitted 2016-11-14; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Intraventricular Haemorrhage Neonatal
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acetaminophen group (Experimental): Babies who took acetaminophen
  Interventions: Drug: Acetaminophen
- Placebo group (Dextrose 5) (Experimental): Babies who took placebo
  Interventions: Drug: Dextrose 5

INTERVENTIONS:
Drug: Acetaminophen — The first group will receive acetaminophen as the following
  1. Loading dose: 20 mg/kg in the first 12-24 hours To be diluted in D5W up to 3-5 ml and to be infused over 15 minutes.
  2. Maintenance dose: 7.5 mg/kg after 6 hrs from the loading dose and to be repeat every 6 hours for 3 days.
  Other Names: Paracetamol
  Arms: acetaminophen group
Drug: Dextrose 5 — The second group will receive placebo (D5W) as the following
  1. Loading dose: 3-5 ml in the first 12-24 hours To be infused over 15 minutes.
  2. Maintenance dose: 3-5 ml after 6 hrs from the loading dose and to be repeat every 6 hours for 3 days.
  Other Names: Dextrose 5%
  Arms: Placebo group (Dextrose 5)

SUMMARY:
The purpose of this study is to determine whether acetaminophen is effective in prevention or reducing the severity of IVH in premature infants.

DETAILED DESCRIPTION:
It will be a double-blind randomized control trial, single center. The study will include neonates with a gestational age of less than or equal 32 weeks and a birth weight of less than or equal 1500 g, and will randomly assigned to two treatment groups (see below).

Infants will be randomized to equal-sized groups using block randomization with blocks of four. Stratified randomization for gender and gestational age will be included in the randomized blocks. Gestational age will be divided into two categories: 23 weeks +0 day to 27 weeks +6 days, and from 28 weeks +0 day to 32 weeks +6 days. Gender (2) × gestational age (2) will give 6 strata, requiring 6 separate random number lists to achieve randomization.

ELIGIBILITY:
Inclusion Criteria:

* Premature baby less than or equal 32 week and birth weight less than or equal 1500 g

Exclusion Criteria:

* Out-born babies, infants with major congenital anomalies, babies have IVH III, IV, High expectancy of early death

Ages: 1 Hour to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of intraventricular hemorrhage (IVH will be graded by Papile score) among the infants on acetaminophen compared to the infants on placebo. | within the first week of age

SECONDARY OUTCOMES:
The incidence of neonatal sepsis in the premature babies who received acetaminophen | Corrected 40 weeks of gestational age or time of discharge will be used
The incidence of Necrotizing Enterocolitis (NEC) in the premature babies who received acetaminophen | Corrected 40 weeks of gestational age or time of discharge will be used
The incidence of bronchopulmonary dysplasia (BPD) in the premature babies who received acetaminophen | Corrected 40 weeks of gestational age or time of discharge will be used

CONTACTS AND LOCATIONS:
Overall Officials: Mountasser Al-Mouqdad, MD, Principal Investigator — King Saud Medical City
Locations (1):
- Mountasser Al-Mouqdad, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No